CLINICAL TRIAL: NCT02580396
Title: Evaluation Of CanADVICE+®M-Health System To Support Breast Cancer Patients Receiving Capecitabine
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Royal Marsden NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CCR4404
Record Dates: First submitted 2015-09-18; First posted 2015-10-20 (Estimated); Last update posted 2018-11-02 (Actual); Status verified 2018-10

CONDITIONS: Metastatic Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Patients eligible for CanADVICE+® (smart phone app) (Other)
  Interventions: Device: CanADVICE+® (smart phone app)

INTERVENTIONS:
Device: CanADVICE+® (smart phone app) — The main objective of this project is to optimise pharmaceutical counselling services by providing drug related information, in a digital format, to patients with metastatic breast cancer receiving Capecitabine.

SUMMARY:
This feasibility study will be conducted in order to provide proof of concept for the CanADVICE+® system comprising a smart phone app and a healthcare organization server side application based on Web 2 technologies. The main objective of this project is to optimise pharmaceutical counselling services by providing drug related information, in a digital format, to patients with metastatic breast cancer receiving Capecitabine.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with metastatic breast cancer
* Commencing first cycle of Capecitabine
* Familiar with and own an android smartphone
* Willing to participate

Exclusion Criteria:

* Patients <18 years
* Patients taking part in any other trial containing Capecitabine
* Chemotherapy-naïve patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2016-03-16 (Actual); Primary Completion 2018-11-01 (Actual); Study Completion 2018-11-01 (Actual)

PRIMARY OUTCOMES:
Patient acceptability of the app using questionnaire provided when patients attend for their 3rd cycle and quantified using a 5-point Likert scale | 42 days
  The app will be used at cycles 1 and 2 of capecitabine (each cycle is 21 days), and acceptability of the app will be measured using a questionnaire when patients attend hospital for their 3rd cycle of capecitabine.

SECONDARY OUTCOMES:
Health care provider's acceptability of the app using questionnaires | 48 months
  At the end of the study, health care professionals (HCPs) involved in the study will be interviewed using semi-structured interview.
Patients' interactivity with the app will be measured using mobile app and web server functions | 42 days
  The app will be used at cycles 1 and 2 of capecitabine (each cycle is 21 days). During this period the number of patient interactions with the mobile app and health care professionals interactions with the web server functions will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Jillian Noble, Principal Investigator — Royal Marsden NHS Foundation Trust
Locations (1):
- The Royal Marsden NHS Foundation Trust, Sutton, Surrey, United Kingdom